CLINICAL TRIAL: NCT06445413
Title: Tai Chi as a Novel Strategy to Increase Physical Activity Among Adults Pursuing Metabolic and Bariatric Surgery: A Feasibility and Acceptability Study
Brief Title: Tai Chi as a Novel Strategy to Increase Physical Activity Among Adults Pursuing Metabolic and Bariatric Surgery
Acronym: ACHIEVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R-HHC-2023-0177
Record Dates: First submitted 2024-02-26; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tai Chi class (Experimental): Participation in ten weekly group in-person Tai Chi classes
  Interventions: Other: Tai Chi

INTERVENTIONS:
Other: Tai Chi — Ten weekly 60-minute Tai Chi classes

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility and acceptability of a 10-wk hybrid Tai Chi (TC) program with in-person classes and online TC videos among 24 physically inactive adults who are seeking metabolic and bariatric surgery (MBS) in a single-arm trial.

The aims are:

Aim 1: Feasibility: To evaluate whether TC is feasible, defined as a mean attendance rate of ≥70% in-person TC classes attended.

Aim 2: Acceptability: To evaluate whether TC is acceptable, defined as a mean rating of ≥4 across 4 acceptability questionnaire items measured on a 5-point Likert scale (e.g., rate "Tai Chi practice is appealing to me" on a scale from 1 [completely disagree] to 5 [completely agree]).

Participants will complete four individual in-person visits where they will complete study assessments and ten weekly group in-person Tai Chi classes where they will practice Tai Chi with up to 5 other study participants. Additionally, they will be asked to practice Tai Chi at home with the aid of instructional online videos and log their practice.

ELIGIBILITY:
Inclusion Criteria:

1. Seeking to undergo MBS at HHC.
2. Be able to give valid informed consent in English. Attending the live, in-person, group TC classes each week is the main component of the intervention. During the classes, the TC instructor will be giving instructions and communicating with the participants in English. It is not practical to having an interpreter during the live classes. Therefore, participation is limited to those who are English speakers.
3. Be 18-70 years of age.
4. Have BMI≥35 kg/m2
5. Absence of cognitive impairment since participants will need to learn and memorize the TC forms. Must score ≥24 Mini-Mental State Examination.
6. Be physically inactive defined as performing <150 min/wk of moderate to vigorous intensity PA based on self-report.
7. Be able to ambulate independently without use of an assistive device.
8. Be able to complete questionnaires and view TC instructional videos via REDCap.
9. Be able to commute to one of the HH Medical and Surgical Weight Loss Center clinics to participate in testing sessions and in-person TC classes.

Exclusion Criteria:

1. Having severe psychological or physical conditions that may impair their ability to adhere to the study protocol such as uncontrolled mental health issues, and severe arthritis.
2. Pregnant women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Attendance | Attendance will be taken at each class (up to 10 weeks)
  Percentage of Tai Chi classes attended over 10 week program
Video view frequency | Measured once weekly for up to 10 weeks
  Number of times the weekly Tai Chi video is viewed
Video view duration | Measured once weekly (up to 10 weeks)
  Number of minutes the weekly Tai Chi video was played
Home practice frequency | Measured once weekly (up to 10 weeks)
  Number of times participant practices Tai Chi at home
Home practice duration | Measured once weekly (up to 10 weeks)
  Number of minutes spent practicing Tai Chi at home
Acceptability of Tai Chi | Measured once at the end of Tai Chi class or when participant drops out
  This is a validated tool to assess the acceptability of interventions with four 5-point Likert scale questions that will be rated from completely disagree to completely agree. Acceptability is defined as a mean rating of ≥4 across 4 acceptability questionnaire items measured on a 5-point Likert scale (e.g., rate "Tai Chi practice is appealing to me" on a scale from 1 [completely disagree] to 5 [completely agree]).

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States